CLINICAL TRIAL: NCT06314425
Title: Prospective Clinical Series With Zirconia Implants
Brief Title: Zirconia Implants: Practice-based Evidence
Acronym: SDS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Dental Solutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB_20240714
Record Dates: First submitted 2024-03-07; First posted 2024-03-18 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Dental Implants; Ceramic Implant
Keywords: ceramic implants; titanium implants; peri-implantitis; marginal bone loss; soft tissue; bone augmentation; immediate implantation; dental implants; immediate loading
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Immediate loading of ceramic implants (Experimental): Tooth/teeth are extracted with minimally invasive approach using piezo surgery and when necessary sectioning after local anesthesia (Articaine 40 mg/mL with epinephrine 10 μg/mL; or Lidocaine 20mg/ml with 10 ug/ml). Extraction sockets are thoroughly degranulated to remove all remnants of soft tissue and residual restorations or material which may have extended beyond the tooth apex. After copious irrigation, the socket condition is recorded, which includes, thickness and location of buccal/facial crestal alveolar bone.
  Interventions: Procedure: Immediate dental implants placements on fresh sockets after tooth extraction

INTERVENTIONS:
Procedure: Immediate dental implants placements on fresh sockets after tooth extraction — Zirconia dental implants (SDS®, Swiss Dental Solution, Kreuzlingen, Switzerland) are to be placed within the fresh extraction sockets. The immediate implants are placed using a minimally invasive technique without vertical releasing incisions. Implant placements are performed following the SDS osteotomy protocol after sulcus marginal and crestal incision or flapless surgery. The same surgeon places implants for all patients. Infected sites are debrided using piezo surgery touch.

SUMMARY:
This study is a prospective case series clinical study to examine the effectiveness of Ceramic dental implants manufactured by Swiss Dental Solutions (SDS). Participants with an indication from the dentist for teeth extraction and replacement are invited to participate in this study. Participating in this study will involve the use of dental implants manufactured by Swiss Dental Solutions (SDS zirconia dental implants), submission of the case data, including pre-operative information, intra-operative details, and post-operative follow-up data, to the study site and its collaborating partners.

The SDS zirconia dental implants used in this research are FDA cleared devices that are available for dental treatments.

DETAILED DESCRIPTION:
To evaluate the effectiveness of one-piece ceramic implants placed into fresh extraction sockets and provide practical clinical evidence, the investigators will assess their performance in defined clinical settings, encompassing a variety of clinical situations, patients, and practitioners. This evaluation, conducted according to a precise surgical and treatment protocol, considers factors such as patient and clinician variability and long-term outcomes in routine clinical practice.

Study Question:

The cumulative survival rate (CSR), Marginal Bone Level (MBL) and Pink Esthetic Score (PES) of one-piece ceramic implants supporting crowns during a 12-month follow-up period will be determined.

ELIGIBILITY:
Inclusion Criteria:

* The need for implant placement in position of single or multiple teeth to be extracted and to replace up to 3 teeth
* Availability of patient for a minimum follow-up of one year following implantation
* Availability of complete follow-up data in medical records
* Availability of post-operative and follow-up periapical radiographs

Exclusion Criteria:

* History of head and neck irradiation
* History of bisphosphonate or medications that induce osteonecrosis of the jaw
* Untreated systemic diseases that are known to affect wound healing, such as uncontrolled diabetes mellitus
* Immunocompromised or immunoproliferative diseases
* Heavy Smoking of >10 cigarettes per day

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-03 (Actual); Primary Completion 2025-04-24 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Cumulative Survival Rate (CSR) | 12-month follow-up
  The cumulative survival rate is determined as the percentage of implants that remained in place over the observation period for each patient. 100% of survival is defined as absence of implant loss.

SECONDARY OUTCOMES:
Marginal Bone Loss (MBL) | 12-month follow-up
  The vertical bone height is measured mesially and distally on intraoral periapical radiographs. The values are assessed at specific time points as follows: T(0) immediately after implant placement, T(1) 6 months after implant placement, T(2) 12 months after implant placement.
  The clinical success of the implants is defined in four groups as follows:
  * Group I < 2 mm of radiographic bone loss without tenderness, mobility, or exudate.
  * Group II radiographic bone loss of 2-4 mm without mobility or tenderness.
  * Group III radiographic bone loss > 4 mm but less than half the implant length with no mobility or exudation.
  * Group IV implant loss.

OTHER OUTCOMES:
Pink Esthetic Score (PES) | 12-month follow-up
  The PES parameters are the presence of papilla (mesial and distal), soft tissue, height of marginal gingiva, alveolar processes, and soft tissue color and texture. The values are assessed at specific time points as follows: T(0) immediately after implant placement, T(1) 6 months after implant placement, T(2) 12 months after implant placement. The seven variables are scored on a scale ranging from 0 to 2 points, with a maximum score of 14 and a minimum score of zero in relation to esthetic parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Etyene Schnurr, DMD PhD DSc MSc, Study Director — Vizstara Professional Education, Clinical and R & D
Locations (1):
- Vizstara Professional Education, Englewood Cliffs, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No